CLINICAL TRIAL: NCT02398656
Title: Multicentre, Prospective Randomized Open Label, Blinded-endpoint (PROBE) Controlled Trial of Thrombolysis With Low Dose Tenecteplase (TNK-tPA) Versus Standard of Care in Minor Ischemic Stroke With Proven Acute Symptomatic Occlusion
Brief Title: A Randomized Controlled Trial of TNK-tPA Versus Standard of Care for Minor Ischemic Stroke With Proven Occlusion
Acronym: TEMPO-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Shelagh B Coutts, Stroke Neurologist, Co- Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version 3.3 , Mar 24,2017
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Stroke, Acute
Keywords: Minor Ischemic Stroke
MeSH Terms: conditions — Stroke | interventions — Tenecteplase; TNK-tissue plasminogen activator; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenecteplase (tNK) (Experimental): Experimental: TNK-tPA (0.25mg/kg) given as a single, intravenous bolus immediately upon randomization. Experimental treatment will be administered as a single intravenous bolus over 1-2 minutes as per the standard manufacturers' instructions for use. Tenecteplase, a genetically engineered mutant tissue plasminogen activator, has a longer half-life, is more fibrin specific, produces less systemic depletion of circulating fibrinogen, and is more resistant to plasminogen activator inhibitor than alteplase.
  Interventions: Drug: Tenecteplase
- Control (Antiplatelet Agents) (Active Comparator): Control: Patients will be treated with standard of care based antiplatelet treatment - choice at the discretion of the investigator. Low dose aspirin (single agent) will be the choice of most physicians, some will chose to use the combination of aspirin and clopidogrel. As this is a multi-centre, international trial where local practices will vary, rather than mandating a specific antiplatelet agent, we will allow the local investigator to chose which antithrombotic regime should be used. Standard of care medication(s) should be given immediately upon randomization.
  Interventions: Drug: Antiplatelet treatment

INTERVENTIONS:
Drug: Tenecteplase — TNK will be administered as a single intravenous bolus over 1-2 minutes within 90 minutes of the CT scan.
  Other Names: TNK-tPA
  Arms: Tenecteplase (tNK)
Drug: Antiplatelet treatment — Low dose aspirin (single agent) will be the choice of most physicians, some Investigators will chose to use the combination of aspirin and clopidogrel.
  Other Names: ASA, Clopidogrel
  Arms: Control (Antiplatelet Agents)

SUMMARY:
This trial will enroll patients that have been diagnosed with a transient ischemic attack (TIA) or minor stroke that has occurred within the past 12 hours. Anyone diagnosed with a minor stroke faces the possibility of long-term disability and even death, regardless of treatment. Stroke symptoms such as weakness, difficulty speaking and paralysis may improve or worsen over the hours or days immediately following a stroke. TEMPO-2 is a minor stroke trial for patients presenting within 12 hours of their symptom onset. Patients will be randomized to TNK-tPA or standard of care. In the intervention group TNK-tPA is given as a single, intravenous bolus (0.25mg/Kg) immediately upon randomization. Maximum dose 50mg. The control group will receive antiplatelet agent(s) as decided by the treating physician. Antiplatelet agent(s) choice will be at the treating physician's discretion.

TEMPO-2 Coordinating Centre is located in Calgary, AB, Canada. There will be approximately 50 sites participating worldwide.

Dr. Shelagh Coutts is the Principal Investigator.

DETAILED DESCRIPTION:
TEMPO2 is an multicentre, prospective randomized open label, blinded-endpoint (PROBE) controlled trial of thrombolysis with low dose Tenecteplase (TNK-tPA) versus standard of care. A total of 1274 patients will be enrolled, at approximately 50 sites worldwide.

TEMPO-2 will enroll patients within a 12 hour time window with a NIHSS score of <6 and an ASPECTS >7. All patients will be evaluated clinically and then undergo brain imaging using CT followed immediately by a CT angiogram. Patients must have an intracranial occlusion on CTA or CTP.

Randomization will be 1:1 to TNK-tPA (experimental) or standard of care antiplatelet agents (control).

Experimental: TNK-tPA (0.25mg/kg) given as a single, intravenous bolus immediately upon randomization. Experimental treatment will be administered as a single intravenous bolus over 1-2 minutes.

Control: Patients will be treated with standard of care based antiplatelet treatment - choice at the discretion of the investigator. Low dose aspirin (single agent) will be the choice of most physicians, some will chose to use the combination of aspirin and clopidogrel. The local investigator to chose which antithrombotic regime should be used

All patients will be treated within 90 minutes of the first slice of the baseline CT. Patients will undergo a study CT angiogram of the intracranial circulation between 4-8 hours after treatment to determine whether the occluded artery has recanalized or not. In sites where MRI/MRA is routinely used this can be substituted for CT/CTA. Any patient who has neurological worsening should have standard of care brain imaging completed to rule out intracranial hemorrhage.

All patients will have standard of care medical management on an acute stroke unit and undergo follow-up imaging at 24 hours with CT or MR. Use of MR will be encouraged.

Patients will be assessed at 24 hours and at Days 5 and 90. The Day 90 Outcomes will be performed by a blinded assessor.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke in an adult patient (18 years of age or older)
2. Onset (last-seen-well) time to treatment time ≤ 12 hours.
3. TIA or minor stroke defined as a baseline NIHSS ≤ 5 at the time of randomization. Patients do not have to have persistent demonstrable neurological deficit on physical neurological examination.
4. Any acute intracranial occlusion or near occlusion (TICI 0 or 1) (MCA, ACA, PCA, VB territories) defined by non-invasive acute imaging (CT angiography or MR angiography) that is neurologically relevant to the presenting symptoms and signs. Multiphase CTA or CT perfusion are required for this study. An acute occlusion is defined as TICI 0 or TICI 1 flow.1 Practically this can include a small amount of forward flow in the presence of a near occlusion AND, Delayed washout of contrast with pial vessels on multiphase CTA in a region of brain concordant with clinical symptoms and signs OR, Any area of focal perfusion abnormality identified using CT or MR perfusion - e.g. transit delay (TTP, MTT or T Max), in a region of brain concordant with clinical symptoms and signs.
5. Pre-stroke independent functional status - structured mRS ≤2.
6. Informed consent from the patient or surrogate.
7. Patients can be treated within 90 minutes of the first slice of CT or MRI. Scans can be repeated to meet this requirement; if there is no change neurologically then only a CT head need be repeated for assessment of extent and depth of ischemia.

Exclusion Criteria:

1. Hyperdensity on NCCT consistent with intracranial hemorrhage.
2. Large acute stroke ASPECTS < 7 visible on baseline CT scan.
3. Core of established infarction. No large area (estimated > 10 cc) of grey matter hypodensity at a similar density to white matter or in the judgment of the enrolling neurologist is consistent with a subacute ischemic stroke > 12 hours of age.
4. Clinical history, past imaging or clinical judgment suggest that that intracranial occlusion is chronic.
5. Patient has a severe or fatal or disabling illness that will prevent improvement or follow-up or such that the treatment would not likely benefit the patient.
6. Pregnancy
7. Planned thrombolysis with IV tPA or endovascular thrombolysis/thrombectomy treatment.
8. In-hospital stroke unless these patients are at their baseline prior to their stroke. E.g. a patient who had a stroke during a diagnostic coronary angiogram.
9. Commonly accepted exclusions for medical thrombolytic treatment. These are commonly relative contraindications (i.e. the final decision is at the discretion of the treating physician) but for the purposes of TEMPO-2 include the following:

   * International normalized ratio > 1.7 or known full anticoagulation with use of any standard or direct oral anticoagulant therapy with full anticoagulant dosing. [DVT prophylaxis dosing shall not prohibit enrolment]. For low molecular weight heparins (LMWH) more than 48 hours off drug will be considered sufficient to allow trial enrollment. For direct oral anticoagulants; in patients with normal renal function more than 48 hours off drug will be considered sufficient to allow trial enrollment. Patients on direct oral anticoagulants who have any degree of renal impairment should not be enrolled in the trial unless they have not taken a dose of the drug in the last 5 days. Dual antiplatelet therapy does not prohibit enrolment.
   * Dual antiplatelet therapy does not prohibit enrolment. [For patients who are known not to be taking anticoagulant therapy it is not necessary to wait for coagulation lab results (e.g. PT, PTT) prior to treatment]
   * Patients who have been acutely treated with GP2b3a inhibitors.
   * Arterial puncture at a non-compressible site in the previous seven days
   * Clinical stroke or serious head or spinal trauma in the preceding three months that would normally preclude use of a thrombolytic agent.
   * History of intracranial hemorrhage, subarachnoid hemorrhage or other brain hemorrhage that would normally preclude use of a thrombolytic agent.
   * Major surgery within the last 3 months at a bodily site where bleeding could result in serious harm or death.
   * Known platelet count below 100,000 per cubic millimeter. Treatment should not be delayed to wait for platelet count unless thrombocytopenia is known or suspected.
   * Gastrointestinal or genitourinary bleeding within the past 3 months that is unresolved or associated with persisting anemia such that thrombolytic treatment of any kind would result in serious bleeding or death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1274 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Hill, MD, Study Director — University of Calgary
Locations (61):
- Australia (7):
  - Calvary Public Hospital Bruce, Canberra, Australian Capital Territory
  - John Hunter Hospital, Newcastle, New South Wales
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (2):
  - Medical University of Vienna (Coordinating Centre), Vienna
  - St. John's of God Hospital Vienna, Vienna
- Brazil (14):
  - Hospital de Clínicas de Botucatu, Botucatu
  - Instituto Hospital de Base do Distrito Federal, Brasília
  - Hospital Universitário Maria Aparecida Pedrossian, Campo Grande
  - Hospital Celso Ramos Florianopolos, Celso Ramos
  - Hospital Geral de Fortaleza, Fortaleza
  - Clinica Neurologica e Neurocirurgica de Joinville Ltda, Joinville
  - Porto Alegre Hospital, Porto Alegre
  - Santa Casa de Porto Alegre, Porto Alegre
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto
  - Americas Medical City, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Hospital São Paulo UNIFESP, São Paulo
  - Irmandade Da Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Hospital Estadual Central, Vitória
- Canada (15):
  - University of Calgary/Foothills Medical Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, B.C.
  - Vancouver General Hospital, Vancouver, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western, Toronto, Ontario
  - McGill University, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - University of Saskatchewan/ Royal University Hospital, Saskatoon, Saskatchewan
- University Central Hospital HUCH, Helsinki, Finland
- Ireland (2):
  - Beaumont Hospital, Dublin, Leinster
  - Mater Misericordiae University Hospital Dublin, Dublin, Leinster
- Christchurch Hospital, Christchurch, New Zealand
- Singapore (2):
  - National Neuroscience Institute Tan Tock Seng Hospital, Singapore
  - Singapore General Hospital, Singapore
- Spain (5):
  - Complejo Jospitalario Universitario A Coruna, A Coruña
  - Vall d'Hebron Institut de Recerca (VHIR), Barcelona
  - Vall d'Hebron Institut de Recerca, Barcelona
  - Hospital Universitari Doctor Josep Trueta, Girona
  - Clinc University Hospital Valladolid, Valladolid
- United Kingdom (12):
  - Countess of Chester, London, England
  - St George's University Hospitals NHS Foundation trust, London, England
  - Stoke University of North Midlands, London, England
  - University College London Hospital, London, England
  - Royal Victoria Hospital, Belfast, Northern Ireland
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrooke Hospital, Cambridge
  - Charring Cross Hospital, London
  - Kings College Hospital, London
  - Nottingham University Hospital, Nottingham
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No
Overall data will be shared once the trial has been closed and data analysed. No individual participant data will be available.

REFERENCES:
- [Result] Coutts SB, Ankolekar S, Appireddy R, Arenillas JF, Assis Z, Bailey P, Barber PA, Bazan R, Buck BH, Butcher KS, Camden MC, Campbell BCV, Casaubon LK, Catanese L, Chatterjee K, Choi PMC, Clarke B, Dowlatshahi D, Ferrari J, Field TS, Ganesh A, Ghia D, Goyal M, Greisenegger S, Halse O, Horn M, Hunter G, Imoukhuede O, Kelly PJ, Kennedy J, Kenney C, Kleinig TJ, Krishnan K, Lima F, Mandzia JL, Marko M, Martins SO, Medvedev G, Menon BK, Mishra SM, Molina C, Moussaddy A, Muir KW, Parsons MW, Penn AMW, Pille A, Pontes-Neto OM, Roffe C, Serena J, Simister R, Singh N, Spratt N, Strbian D, Tham CH, Wiggam MI, Williams DJ, Willmot MR, Wu T, Yu AYX, Zachariah G, Zafar A, Zerna C, Hill MD; TEMPO-2 investigators. Tenecteplase versus standard of care for minor ischaemic stroke with proven occlusion (TEMPO-2): a randomised, open label, phase 3 superiority trial. Lancet. 2024 Jun 15;403(10444):2597-2605. doi: 10.1016/S0140-6736(24)00921-8. Epub 2024 May 17. PMID 38768626
- [Derived] Zhang Y, Buck BH, Barber PA, Chatterjee K, Clarke B, Choi PMC, Hunter G, Ganesh A, Mishra SM, Williams D, Campbell BCV, Dowlatshahi D, Butcher KS, Krishnan K, Wiggam MI, Kleinig TJ, Muir KW, Zerna C, Field TS, Goyal M, Yu AYX, Roffe C, Demchuck AM, Parsons MW, Bazan R, Ankolekar S, Kennedy J, Menon BK, Mandzia JL, Pille A, Kelly PJ, Marko M, Singh N, Vatanpour S, Lima FO, Catanese L, Horn M, Ghia D, Ferrari J, Greisenegger S, Hill MD, Coutts SB; TEMPO-2 Investigators. Thrombolysis With Tenecteplase for Minor Disabling Stroke: Secondary Analysis of the TEMPO-2 Randomized Clinical Trial. JAMA Neurol. 2025 Dec 1;82(12):1243-1250. doi: 10.1001/jamaneurol.2025.4152. PMID 41143808
- [Derived] Logallo N, Kvistad CE, Thomassen L. Therapeutic Potential of Tenecteplase in the Management of Acute Ischemic Stroke. CNS Drugs. 2015;29(10):811-8. doi: 10.1007/s40263-015-0280-9. PMID 26387127

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tenecteplase (tNK) | Control (Antiplatelet Agents)
Started | 637 | 637
Completed | 454 | 432
Not Completed | 183 | 205

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenecteplase (tNK) | Control (Antiplatelet Agents) | Total
Number analyzed (Participants) | 432 | 452 | 884
Age, Continuous [Mean (Full Range); unit: years] | 72 [62 to 80] | 72 [61 to 79] | 72 [61 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 180 | 368
  Male | 244 | 272 | 516
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 14
  Not Hispanic or Latino | 427 | 443 | 870
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 5 | 9
  Asian | 40 | 42 | 82
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 7 | 13
  White | 371 | 382 | 753
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 16 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Return to Baseline Neurological Functioning Measured by the Modified Rankin Scale (mRS)
Description: Analysis will be a responder analysis where return to baseline level of neurological functioning is defined as follows:
  If pre-morbid mRS is 0-1 then mRS 0-1 at 90 days is a good outcome. If pre-morbid mRS is 2 then mRS 0-2 is a good outcome.
  Pre-morbid mRS is assessed using the structured mRS prior to randomization. Outcomes at 90 days will be assessed by an individual blinded to the treatment assignment. The 90day mRS will be rated using the structured mRS questionnaire . The 90 day mRS will be completed in person where possible and by telephone otherwise. The structured questionnaire has been showed to improve reliability in assessing the mRS both in person and by telephone. This is a scale from 0-6. Higher scores mean a worse outcome.
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (tNK) | Control (Antiplatelet Agents)
Number analyzed (Participants) | 432 | 452
Participants | 309 | 338
Statistical Analysis 1: Comparison: Tenecteplase (tNK) vs Control (Antiplatelet Agents); Test type: Superiority; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.88 to 1.04]

2. Secondary Outcome: Number of Participants With Modified Rankin Score (mRS) 0-1 at 90 Days
Description: Pre-morbid mRS is assessed using the structured mRS prior to randomization. Outcomes will be assessed by an individual blinded to the treatment assignment. The 90day mRS will be rated using the structured mRS questionnaire . The 90 day mRS will be completed in person where possible and by telephone otherwise. The structured questionnaire has been showed to improve reliability in assessing the mRS both in person and by telephone. This is a scale from 0-6. Higher scores mean a worse outcome.
  mRS 0-1 represents excellent functional outcome.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (tNK) | Control (Antiplatelet Agents)
Number analyzed (Participants) | 432 | 452
Participants | 298 | 321

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization to Day 5 or discharge ( whichever was sooner). SAE's were collected to the Day 90 assessment completion. AEs and SAE's were collected from the beginning of the trial until the last Day 90 assessment was completed.
Description: AE and SAE definitions are as per GCP requirements.
Arm/Group | Tenecteplase (tNK) | Control (Antiplatelet Agents)
All-Cause Mortality (participants affected / at risk) | 20/425 | 5/442
Serious Adverse Events (participants affected / at risk) | 16/432 | 2/452
Other Adverse Events (participants affected / at risk) | 35/435 | 33/452
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenecteplase (tNK) (N=432) | Control (Antiplatelet Agents) (N=452)
Symptomatic Intracerebral hemorrhage (Nervous system disorders) | 16 (16) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenecteplase (tNK) (N=435) | Control (Antiplatelet Agents) (N=452)
Stroke Progression (Nervous system disorders) | 35 (35) | 33 (33)

LIMITATIONS AND CAVEATS:
The trial was ended based on a recommendation from the DSMB that to continue was futile.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT02398656/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT02398656/SAP_001.pdf